CLINICAL TRIAL: NCT05386433
Title: The Effect of Paxlovid in the Treatment of COVID-19 Patients With Uremia
Brief Title: Paxlovid in the Treatment of COVID-19 Patients With Uremia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, PhD, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PaxlovidUremia
Record Dates: First submitted 2022-05-20; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Uremia
MeSH Terms: conditions — COVID-19; Uremia | interventions — nirmatrelvir and ritonavir drug combination; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard-of-care (Placebo Comparator): Standard-of-care of COVID-19 includes oxygen inhalation, antibiotics, traditional medicine, etc.
  Interventions: Drug: standard-of-care
- standard-of-care plus Paxlovid (Experimental): standard-of-care of COVID-19 plus Paxlovid
  Interventions: Drug: Paxlovid; Drug: standard-of-care

INTERVENTIONS:
Drug: Paxlovid — Paxlovid contains two medicines: nirmatrelvir and ritonavir. Nirmatrelvir [PF-07321332] is a SARS-CoV-2 main protease (Mpro) inhibitor (also known as SARS-CoV2 3CL protease inhibitor) that works by inhibiting viral replication in the early stages of the disease to prevent progression to severe COVID-19.
  Ritonavir is co-administered with nirmatrelvir to help slow its metabolism in order for it to remain active in the body for longer periods of time at higher concentrations to help combat the virus.
  Arms: standard-of-care plus Paxlovid
Drug: standard-of-care — standard-of-care of COVID-19

SUMMARY:
This study is a single-center, open-label, randomized controlled clinical study to evaluate the effect of Paxlovid on the virus-negative time and disease progression in uremic patients infected with SARS-CoV-2 (omicron variants).

This study will enroll maintenance hemodialysis patients infected with SARS-CoV-2 (omicron variants).

After signing the informed consent form, the qualified subjects will be randomly stratified 1:1 to standard-of-care (SOC) or SOC plus Paxlovid for five days.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent. Age ≥ 18 years old. COVID-19 (nucleic acid test positive) was diagnosed before randomization. At least 1 symptom or sign of COVID-19 at the time of being enrolled into the study(symptoms and signs related to COVID-19 including cough, expectoration, dyspnea, fever, chills, fatigue, muscle soreness, diarrhea, headache, sore throat, stuffy nose, runny nose, etc.).

Exclusion Criteria:

* History of active liver disease, including chronic or active hepatitis B or C, primary biliary cirrhosis, Child-Pugh B or C, or acute liver failure.

HIV infection and the viral load is greater than 400 copies/ml. Suspected or confirmed active systemic infections that may have an impact on the study evaluation except for COVID-19.

Acute heart failure, respiratory failure, severe chronic kidney disease, and cardiovascular disease caused by uremia-related complications.

Allergic to any ingredients of Paxlovid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
time of negative conversion of SARS-CoV-2 nucleic acid | up to 60 days
  Time from first positive to negative of SARS-CoV-2 nucleic acid
Proportion of ICU transfer or disease progression to severe or critical illness | up to 60 days

IPD SHARING:
Plan to Share IPD: No